CLINICAL TRIAL: NCT00936195
Title: Safety and Efficacy of the Universal Use of EFV-TDF-FTC and AZT-3TC-LPV/r Combinations in Pregnant and Breastfeeding Women to Prevent mother-to Child Transmission of HIV-1 o, Resource-limited Settings: A Multicentre Randomized Phase 3 Clinical Trial
Brief Title: Universal Use of EFV-TDF-FTC and AZT-3TC-LPV/r Combinations for HIV-1 PMTCT in Pregnant and Breastfeeding Women : a Phase 3 Trial
Acronym: UMA
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: faillure to obtain insurance because of refusal from insurance companies
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: Gilead Sciences (Industry); Merck Sharp & Dohme LLC (Industry); GlaxoSmithKline (Industry); Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ANRS 12200 UMA
Record Dates: First submitted 2009-07-08; First posted 2009-07-09 (Estimated); Last update posted 2012-02-15 (Estimated); Status verified 2012-02

CONDITIONS: HIV Infection; Pregnancy; Breastfeeding; HIV Infections
Keywords: HIV; pregnancy; breastfeeding; PMTCT; ARV treatment; treatment naive
MeSH Terms: conditions — HIV Infections; Breast Feeding | interventions — Efavirenz, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atripla (R) (Active Comparator)
  Interventions: Drug: Efavirenz-Tenofovir-Emtricitabine
- Combivir (R) + Kaletra (R) or Aluvia (R) (Active Comparator)
  Interventions: Drug: Zidovudine-Lamivudine-Lopinavir/Ritonavir

INTERVENTIONS:
Drug: Efavirenz-Tenofovir-Emtricitabine — Atripla (R) : Efavirenz 600 mg - Tenofovir 300 mg - Emtricitabine 200 mg; Dosage : 1 pill/day
  Arms: Atripla (R)
Drug: Zidovudine-Lamivudine-Lopinavir/Ritonavir — Combivir (R) : Zidovudine 300 mg - Lamivudine 150 mg Dosage : 1 pill twice a day
  Kaletra (R) or Aluvia (R) : Lopinavir 200 mg / Ritonavir 50 mg Dosage : 2 or 3 pills twice a day
  Arms: Combivir (R) + Kaletra (R) or Aluvia (R)

SUMMARY:
To assess the maternal and infant safety of a single daily fixed-dose combination of TDF/FTC/EFV (Atripla®), compared to the association of LPV/r (Kaletra® or Aluvia®) and 3TC/ZDV (Combivir®) given to African women to prevent overall MTCT in populations practicing breastfeeding.

DETAILED DESCRIPTION:
The prevention of MTCT during pregnancy and through breastfeeding exposure remains challenging to date in most resource-limited settings. Peripartum HIV transmission is already amenable to ARV interventions. These ARV regimens, partially efficacious are insufficiently used despite their apparent simplicity. The postnatal transmission via breastfeeding remains a serious additional threat.

This is a multicentric, non-inferiority, randomized controlled trial aiming at assessing the maternal and infant safety of a single daily fixed-dose combination of TDF/FTC/EFV (Atripla®), compared to the association of LPV/r (Kaletra® or Aluvia®) and 3TC/ZDV (Combivir®) given to African women (in Cote d'Ivoire an in Zambia) to prevent MTCT overall in breastfeeding population.

The fixed-dose combination of Tenofovir/Emtricitabine/Efavirenz (TDF/FTC/EFV or Atripla®) is a highly effective HAART combination and the simplest ARV regimen currently available in resource-limited settings and is therefore likely to become soon the lead first-line HAART regimen for adults in such settings. Its anticipated widespread prescription in women of childbearing age requires the proper documentation of its use in pregnancy and during breastfeeding.

The combination of ZDV/3TC (Combivir®) and Lopinavir/ritonavir (LPV/r) (Kaletra® or Aluvia®) is chosen as a reference regimen as it is one of the most commonly used first-line HAART for adults and the reference regimen for PMTCT in industrialised settings.

The maternal ARV regimen will be initiated as soon as possible from 20 weeks of gestation until at least the cessation of breastfeeding (with the advice to cease at six months). The decision to stop or continue the maternal ARV regimen after breastfeeding cessation will be based on the baseline maternal CD4 count and the maternal clinical stage at baseline and/or at breastfeeding cessation. A woman with a baseline CD4 <500 cells/ml will always be proposed to continue her treatment after breastfeeding cessation. A woman with a baseline CD4 count >500 will be asked to stop her treatment after breastfeeding cessation unless she has reached the WHO clinical stage IV at that time.

Infants will receive daily Zidovudine syrup from birth during the first week of life, or an updated ARV post-exposure prophylaxis recommended by WHO when women receive HAART.

ELIGIBILITY:
Inclusion Criteria:

* being pregnant, presenting in at least the 20th week of pregnancy and no later than 2 weeks before the expected term;
* at least 18 years of age;
* diagnosed as infected with HIV-1 only;
* not currently taking any ARV drugs;
* having not been exposed to NVP in the 6 months preceding enrolment;
* willing to breastfeed their forthcoming child;
* residing and planning to continue to reside within the predefined catchment areas until 12 months after delivery;
* being able to give informed consent for enrolment in the study;
* lacking any medical contraindication to any of the proposed ARV medications;
* and accepting the principle of being randomized to receive one of the ARV regimens evaluated within the study, to prevent MTCT and for their own health when required.

Exclusion Criteria:

* presenting within 2 weeks before the expected term;
* currently taking ARV drugs;
* having been exposed to NVP in the 6 months preceding enrolment;
* not willing to breastfeed their forthcoming child;
* having severe renal insufficiency (creatin clearance < 60ml/min);
* diagnosed as infected with HIV-2 only or dually infected HIV-1 and HIV-2;
* hemoglobin < 7 g/dL in the month preceding inclusion
* HBs Ag positive

Women meeting one of the three last exclusion criteria (HIV-2 infection or co-infection, hemoglobin < 7 g/dL, HBs Ag positive) will not be randomized but will all received Atripla and be followed-up in an ancillary open cohort according the same procedures and agenda.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-01; Primary Completion 2013-01 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
cumulative occurence of : -adverse pregnancy outcomes (spontaneous abortion, stillbirth, congenital abnormality requiring surgical correction in children < 1 yr of age); -paediatric HIV infection; -infant mortality | at 6 and 12 months following delivery/birth

SECONDARY OUTCOMES:
occurence of grade 4 events in treated women, and of grade 3 or 4 events in ARV-exposed infants | at 6 and 12 months following delivery/birth
frequency of virological failure (>300 copies/mL) and viral resistance profile | at 6 month and 12 months post-delivery
frequency of premature delivery (<37 weeks) and frequency of low birth weight (<2500 g) | at delivery/birth
cumulative incidence of paediatric HIV infection | at 12 months after delivery
tolerability of the ARV combination in treated women | at 6 and 12 months following delivery/birth

CONTACTS AND LOCATIONS:
Overall Officials: Didier K Ekouevi, MD, PhD, Study Chair — Programme PACCI Abidjan, Cote d'Ivoire; François Dabis, MD, PhD, Study Chair — Bordeaux 2 University, France
Locations (2):
- Programme PAC-CI, site ANRS, Abidjan, Côte d’Ivoire
- Center for Infectious Desease Reserach in Zambia, Lusaka, Zambia